CLINICAL TRIAL: NCT04053075
Title: Cluster Linkage Using Statistics to Trigger and Evaluate Response (CLUSTER) Trial for Outbreak Detection and Response
Brief Title: CLUSTER Trial for Outbreak Detection and Response
Acronym: CLUSTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Hospital Corporation of America (Industry); Brigham and Women's Hospital (Other); University of California, Irvine (Other); Harvard School of Public Health (HSPH) (Other); Rush University (Other); Duke University (Other); University of Massachusetts, Amherst (Other); University of California, San Francisco (Other); Cook County Health & Hospitals System (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Platt, Professor and Department Chair, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PH000599B
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Cluster Detection
Keywords: Hospital Outbreak Detection; Hospital Outbreak Response; Cluster; Multidrug Resistant Organism; Genetic Relatedness; Whole Genome Sequencing

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine cluster detection (Active Comparator): Hospitals will use routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Interventions: Other: Routine cluster detection
- Enhanced cluster detection (Active Comparator): Hospitals will use an automated statistical cluster detection tool in addition to routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Interventions: Other: Enhanced cluster detection

INTERVENTIONS:
Other: Routine cluster detection — Hospitals will use routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Arms: Routine cluster detection
Other: Enhanced cluster detection — Hospitals will use an automated statistical cluster detection tool in addition to routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Arms: Enhanced cluster detection

SUMMARY:
Despite the critical importance of identifying hospital-associated outbreaks as early as possible in order to limit their spread, there are currently no standardized methods for cluster detection. The CLUSTER Trial (Cluster Linkage Using Statistics to Trigger and Evaluate Response) will assess whether a statistically-based automated cluster detection method coupled with a robust response protocol will enable rapid containment of hospital clusters as measured by a reduction in cluster size and duration as compared to routine hospital cluster detection methods coupled with the same response protocol.

Note: that enrolled "subjects" represents 82 individual HCA Healthcare hospitals that have been randomized

ELIGIBILITY:
Facility Inclusion Criteria:

* All U.S. HCA Healthcare hospitals that provide inpatient care.
* Facilities that are reporting to the centralized data warehouse during the study period.

Facility Exclusion Criteria:

-

Note: unit of randomization is the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2905455 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Platt, MD, MSc, Principal Investigator — Harvard Pilgrim Health Care Institute; Susan Huang, MD, MPH, Principal Investigator — University of California, Irvine; Meghan Baker, MD, ScD, Study Director — Brigham and Women's Hospital
Locations (82):
- United States (82):
  - Riverside Community Hospital, Riverside, California
  - Regional Medical Center of San Jose, San Jose, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Swedish Medical Center, Denver, Colorado
  - Sky Ridge Medical Center, Denver, Colorado
  - Presbyterian St. Luke's Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - North Suburban Medical Center - JV, Thornton, Colorado
  - JFK Medical Center, Atlantis, Florida
  - Brandon Regional, Brandon, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Lake City Medical Center, Lake City, Florida
  - Largo Medical Center, Largo, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - West Marion Community Hospital, Ocala, Florida
  - Raulerson Hospital, Okeechobee, Florida
  - Orange Park Medical Center, Orange Park, Florida
  - Gulf Coast Medical Center, Panama City, Florida
  - West Florida Hospital, Pensacola, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - St. Lucie Medical Center, Port Saint Lucie, Florida
  - Central Florida Regional Hospital, Sanford, Florida
  - Doctor's Hospital Sarasota, Sarasota, Florida
  - Northside Hospital, St. Petersburg, Florida
  - South Bay Hospital, Sun City Center, Florida
  - Medical Center of Trinity, Trinity, Florida
  - JFK Medical Center - North Campus, West Palm Beach, Florida
  - Fairview Park, Dublin, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Eastside Medical Center, Snellville, Georgia
  - West Valley Medical Center, Caldwell, Idaho
  - Eastern Idaho Regional, Idaho Falls, Idaho
  - Menorah Medical Center, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wesley Woodlawn Hospital, Wichita, Kansas
  - Greenview Regional Hospital, Bowling Green, Kentucky
  - Garden Park Medical Center, Gulfport, Mississippi
  - Research Medical Center, Kansas City, Missouri
  - Lee's Summit Medical Center, Lee's Summit, Missouri
  - Mountainview Hospital - Vegas, Las Vegas, Nevada
  - Parkland Medical Center, Derry, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Spotsylvania Regional Medical Center, Fredericksburg, Pennsylvania
  - Trident Regional Medical Center, Charleston, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Summerville Medical Center, Summerville, South Carolina
  - Colleton Medical Center, Walterboro, South Carolina
  - TriStar Horizon Medical Center, Dickson, Tennessee
  - Summit Medical Center, Hermitage, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Southern Hills Medical Center, Nashville, Tennessee
  - Medical City Arlington, Arlington, Texas
  - St. David's Medical Center, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - Conroe Regional Medical Center, Conroe, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Medical City Denton, Denton, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - Medical City Alliance, Fort Worth, Texas
  - St. David's Georgetown Hospital, Georgetown, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Medical Center of Lewisville, Lewisville, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - Medical City McKinney, McKinney, Texas
  - Medical City North Hills, North Richland Hills, Texas
  - Methodist Hospital, San Antonio, Texas
  - Methodist Stone Oak Hospital, San Antonio, Texas
  - Northeast Methodist Hospital, San Antonio, Texas
  - Mainland Medical Center, Texas City, Texas
  - Clearlake Regional Medical Center, Webster, Texas
  - Ogden Regional Medical Center, Ogden, Utah
  - LewisGale Hospital - Montgomery, Blacksburg, Virginia
  - Reston Hospital, Reston, Virginia
  - Retreat Doctors' Hospital, Richmond, Virginia
  - CJW Medical Center (Chippenham Campus), Richmond, Virginia
  - CJW Medical Center (Johnston Willis Campus), Richmond, Virginia
  - Henrico Doctors' Hospital - Forest Campus, Richmond, Virginia
  - Henrico Doctors' Hospital - Parham Campus, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baker MA, Septimus E, Kleinman K, Moody J, Sands KE, Varma N, Isaacs A, McLean LE, Coady MH, Blanchard EJ, Poland RE, Yokoe DS, Stelling J, Haffenreffer K, Clark A, Avery TR, Sljivo S, Weinstein RA, Smith KN, Carver B, Meador B, Lin MY, Lewis SS, Washington C, Bhattarai M, Shimelman L, Kulldorff M, Reddy SC, Jernigan JA, Perlin JB, Platt R, Huang SS. A Trial of Automated Outbreak Detection to Reduce Hospital Pathogen Spread. NEJM Evid. 2024 May;3(5):EVIDoa2300342. doi: 10.1056/EVIDoa2300342. Epub 2024 Apr 23. PMID 38815164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 out of 182 HCA Healthcare hospitals were recruited for this trial. There was a 30 month intervention period from July 2019 through January 2022.
Pre-assignment Details: 2,905,455 patients were involved in the intervention period from the 82 participating hospitals.
Units Other Than Participants: Hospitals
Period: Overall Study
Arm/Group | Routine Cluster Detection | Enhanced Cluster Detection
Started | 1446854; 41 Hospitals | 1458601; 41 Hospitals
Completed | 1446854; 39 Hospitals | 1458601; 40 Hospitals
Not Completed | 0; 2 Hospitals | 0; 1 Hospitals

BASELINE CHARACTERISTICS:
Population: Number of participant totals reflect total Intervention participants. 82 hospitals were randomized to a study group, 41 began the assigned intervention. 1 hospital withdrew from the intervention arm and 2 hospitals withdrew from the control arm.
Groups:
- Arm 1: Routine Cluster Detection: Hospitals will use routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Routine cluster detection: Hospitals will use routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
- Arm 2: Enhanced Cluster Detection: Hospitals will use an automated statistical cluster detection tool in addition to routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
  Enhanced cluster detection: Hospitals will use an automated statistical cluster detection tool in addition to routine practices for cluster detection with a structured cluster response protocol when a cluster is detected.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Routine Cluster Detection | Arm 2: Enhanced Cluster Detection | Total
Number analyzed (Participants) | 1446854 | 1458601 | 2905455
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.0 [32.0 to 73.0] | 56.0 [32.0 to 72.0] | 57.0 [32.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    number analyzed (Participants) | 1443661 | 1454501 | 2898162
    Female | 800932 | 805509 | 1606441
    Male | 642729 | 648992 | 1291721
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1017301 | 996468 | 2013769
  Race: Black | 196654 | 229501 | 426155
  Race: Other | 84017 | 65406 | 149423
  Race: Unknown | 148882 | 167226 | 316108

OUTCOME MEASURES:

1. Primary Outcome: Cluster Size
Description: Cluster size defined as number of cases identified after the initial cluster signal through the last cluster case.
  NOTE: this outcome is intended for the primary manuscript.
Time Frame: 30 months
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number (95% Confidence Interval); unit: outbreak cases after first signal
Arm/Group | Arm 1: Routine Cluster Detection | Arm 2: Enhanced Cluster Detection
Number analyzed (Participants) | 1446854 | 1458601
outbreak cases after first signal | 1.81 [1.11 to 2.96] | 1.41 [0.88 to 2.24]

2. Secondary Outcome: Cluster Duration
Description: Cluster duration defined as number of days from the initial cluster signal through the last cluster case.
  NOTE: this outcome is intended for the primary manuscript.
Time Frame: 30 months
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Arm 1: Routine Cluster Detection | Arm 2: Enhanced Cluster Detection
Number analyzed (Participants) | 1446854 | 1458601
days | 1.12 [0.81 to 1.56] | 0.88 [0.64 to 1.21]

3. Other Pre Specified Outcome: Genetic Relatedness of Clusters of Microbial Isolates
Description: Compare the genetic relatedness of isolates within a cluster, defined by the automated cluster detection tool or routine cluster detection methods.
  NOTE: this exploratory analysis is intended for a secondary manuscript.
Time Frame: 30 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Pathogen Subgroup Analysis
Description: Subset analyses of trial outcomes (e.g., Gram-positive clusters, Gram-negative clusters, fungal clusters, Clostridium difficile & multidrug-resistant organism clusters).
  NOTE: this exploratory analysis is intended for a secondary manuscript.
Time Frame: 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 Months
Arm/Group | Arm 1: Routine Cluster Detection | Arm 2: Enhanced Cluster Detection
All-Cause Mortality (participants affected / at risk) | 0/1446854 | 0/1458601
Serious Adverse Events (participants affected / at risk) | 0/1446854 | 0/1458601
Other Adverse Events (participants affected / at risk) | 0/1446854 | 0/1458601

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT04053075/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04053075/SAP_001.pdf